CLINICAL TRIAL: NCT02741219
Title: A Multicenter Study: Dexmedetomidine Combined With Sufentanil for Patient Controlled Intravenous Analgesia After Caesarean Section
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Obstetrics & Gynecology Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Nie Yuyan, Associate Professor, Obstetrics & Gynecology Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OBGynFudanU
Record Dates: First submitted 2016-03-11; First posted 2016-04-18 (Estimated); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Saline Solution; Dexmedetomidine; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- Control Group (Placebo Comparator): Parturients in this group receive 20ml intravenous normal saline immediately after delivery. Their patient controlled analgesia (PCA) protocol after surgery consists of 100 mcg sufentanil diluted into 100ml and administer at a background infusion of 1ml/h,and a bolus of 2ml, with a lock-out of 8min.
  Interventions: Drug: Normal saline; Drug: Sufentanil
- Dex Group (Experimental): Parturients in this group receive 0.5mcg/kg intravenous dexmedetomidine diluted to 20ml with normal saline. Their PCA protocol after surgery is 100mcg sufentanil and 300mcg dexmedetomidine diluted to 100ml in saline, with the continuous infusion of 1ml/h, and a bolus of 2 ml, with a lock-out of 8min.
  Interventions: Drug: Dexmedetomidine; Drug: Sufentanil and dexmedetomidine

INTERVENTIONS:
Drug: Normal saline — Control Group receives normal saline bolus after delivery
  Arms: Control Group
Drug: Dexmedetomidine — Dex Group receives dexmedetomidine bolus 0.5mcg/kg after delivery
  Arms: Dex Group
Drug: Sufentanil — sufentanil PCA after surgery
  Arms: Control Group
Drug: Sufentanil and dexmedetomidine — sufentanil combined with dexmedetomidine PCA after surgery
  Arms: Dex Group

SUMMARY:
The purpose of this multicenter study is to evaluate the effectiveness and safety of dexmedetomidine combined with sufentanil for patient-controlled analgesia after caesarean section

ELIGIBILITY:
Inclusion Criteria:

1. Parturients undergoing elective caesarean delivery under spinal anaesthesia
2. American Society of Anesthesiologists class I and II parturients aged 18-45 years, with term singleton pregnancies
3. Parturients with the ability to understand verbal and written mandarin
4. Parturients who want to use PCA intravenous analgesia and can use the pump correctly
5. Parturients whose written informed consent have been obtained

Exclusion Criteria:

1. A history of allergy to dexmedetomidine or other study drugs
2. A long use history of opioid analgesic, NSAIDs, tranquilliser use
3. Psychiatric disorders
4. A history of neuromuscular and endocrine disease or allergic disease
5. A history of lower abdominal surgery
6. Preoperative heart rate (HR) less than 50 bpm, SBP less than 100 mmHg or cardiac conduction or rhythm abnormalities
7. spinal anaesthesia was unsuccessful or an epidural catheter had to be used to achieve adequate anaesthesia
8. A second operation is required during the study.
9. Participating other study during the latest three months
10. Body mass index more than 30 kg/m2
11. Difficult airway ( Mallampati score more than 3 and anatomic deformity )
12. Not suitable for participation estimated by investigation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 225 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Sufentanil consumption | During 24h after surgery
  The total consumption of sufentanil during 24h after surgery are recorded.
Changes in pain score | At 0, 4, 8 and 24 h after surgery
  Pain scores at rest and movement are evaluated with a visual analogue scale (VAS).

SECONDARY OUTCOMES:
Changes in Ramsay sedation score (RSS) | At 4, 8 and 24 h after surgery
  Sedation intensity measured with RSS is recorded at the 4, 8 and 24 h after surgery.
Changes in systolic blood pressure | At 0 min, 5 min, 10 min, 30 min after intervention during surgery and at 8h,24 h after surgery.
  Systolic blood pressure is recorded at 0 min, 5 min, 10 min, 30 min after intervention during surgery and at 8h,24 h after surgery.
Press times of analgesic pump | During 24h after surgery
  The total press times and invalid press times are recorded during 24h after surgery.
Changes in heart rate (HR) | At 0 min, 5 min, 10 min, 30 min after intervention during surgery and at 8h,24 h after surgery
  HR is recorded at 0 min, 5 min, 10 min, 30 min after intervention during surgery and at 8h,24 h after surgery.
Changes in saturation of blood oxygen (SpO2) | At 0 min, 5 min, 10 min, 30 min after intervention during surgery and at 8h,24 h after surgery
  SpO2 is recorded at 0 min, 5 min, 10 min, 30 min after intervention during surgery
Changes in diastolic blood pressure | At 0 min, 5 min, 10 min, 30 min after intervention during surgery and at 8h,24 h after surgery
  Diastolic blood pressure is recorded at 0 min, 5 min, 10 min, 30 min after intervention during surgery and at 8h,24 h after surgery.
Changes in mean arterial blood | At 0 min, 5 min, 10 min, 30 min after intervention during surgery and at 8h,24 h after surgery
  Mean arterial blood pressure is recorded at 0 min, 5 min, 10 min, 30 min after intervention during surgery and at 8h,24 h after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Obstetrics & Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality, China